CLINICAL TRIAL: NCT02639637
Title: Contribution of Neuropeptide Y (NPY) to Vasoconstriction and Sympathetic Activation in the Setting of Dipeptidyl Peptidase IV (DPP4) Inhibition
Brief Title: Effect of DPP4 Inhibition on Vasoconstriction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, MD, Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 151133
Record Dates: First submitted 2015-12-16; First posted 2015-12-24 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Sitagliptin; Dipeptidyl Peptidase IV Inhibitors; Angiotensin Converting Enzyme Inhibitors; Enalaprilat; Neuropeptide Y
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; microcrystalline cellulose; Neuropeptide Y; Enalaprilat; Valsartan

STUDY DESIGN:
Intervention Model Description: Crossover Arms 1 and 2, Crossover Arms 3 and 4
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sitagliptin then Placebo (Other): Subjects in this arm will receive sitagliptin 100 mg daily. After one week of treatment, subjects will report for study day #1. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. A four week washout of medications will occur after the study day. Subjects will then receive placebo for one week followed by study day #2.
  Interventions: Drug: Sitagliptin; Drug: Placebo; Drug: Neuropeptide Y; Drug: Enalaprilat
- Placebo then Sitagliptin (Other): Subjects in this arm will receive placebo for one week. After this, subjects will report for study day #1. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. A four week washout of medications will occur after the study day. Subjects will then receive 100 mg of sitagliptin daily for one week followed by study day #2.
  Interventions: Drug: Sitagliptin; Drug: Placebo; Drug: Neuropeptide Y; Drug: Enalaprilat
- Sitagliptin then Placebo: Valsartan (Placebo Comparator): Subjects in this arm will receive sitagliptin 100 mg/d for one week as well as valsartan 160 mg/d for one week. After this subjects will report for study day #1. During the study day, subjects will be given intra-arterial neuropeptide Y. A four week washout of medication will occur after the study day. Subjects will then receive placebo/d and valsartan 160 mg/d for one week followed by study day #2.
  Interventions: Drug: Sitagliptin; Drug: Placebo; Drug: Valsartan 160mg
- Placebo then Sitagliptin: Valsartan (Placebo Comparator): Subjects in this arm will receive placebo/d for one week as well as valsartan 160 mg/d for one week. After this subjects will report for study day #1. During the study day, subjects will be given intra-arterial neuropeptide Y. A four week washout of medication will occur after the study day. Subjects will then receive sitagliptin 100mg/d and valsartan 160 mg/d for one week followed by study day #2.
  Interventions: Drug: Sitagliptin; Drug: Placebo; Drug: Valsartan 160mg

INTERVENTIONS:
Drug: Sitagliptin — Subjects will receive sitagliptin 100 mg daily for 7 days prior to one of the study days.
  Other Names: Januvia
Drug: Placebo — Subjects will receive a placebo capsule daily for 7 days prior to one of the study days.
  Other Names: Microcrystalline cellulose
Drug: Neuropeptide Y — During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Other Names: NPY
  Arms: Placebo then Sitagliptin; Sitagliptin then Placebo
Drug: Enalaprilat — Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second infusion of neuropeptide Y will begin. Similar to the previous neuropeptide infusion, four doses of neuropeptide Y will be used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Other Names: Vasotec I.V.
  Arms: Placebo then Sitagliptin; Sitagliptin then Placebo
Drug: Valsartan 160mg — Valsartan 160 mg/d for 7 days prior to one of the study days.
  Other Names: valsartan p.o.
  Arms: Placebo then Sitagliptin: Valsartan; Sitagliptin then Placebo: Valsartan

SUMMARY:
The purpose of this study is to understand how dipeptidyl peptidase IV (DPP4) inhibition in diabetics affects hemodynamic parameters and sympathetic activation in the setting of increasing concentrations of neuropeptide Y, an endogenous peptide. The central hypothesis is that DPP4 inhibition decreases degradation of neuropeptide Y, resulting in increased vasoconstriction and sympathetic activation.

DETAILED DESCRIPTION:
Dipeptidyl peptidase IV (DPP4) inhibitors are routinely used for the treatment of type II diabetes mellitus (T2DM). Since the prevalence of hypertension is 1.5-3 times greater in diabetics compared to sex-aged matched controls, the use of antihypertensives such as ACE inhibitors is also common in diabetics. DPP4 is involved in the degradation of multiple vasoactive peptides, one of which is neuropeptide Y. This peptide is thought to play a role in blood pressure regulation and sympathetic nervous system activation. The aim of this study is to investigate how DPP4 inhibition affects vasoconstriction in response to increasing neuropeptide Y concentrations. Additionally, the investigators want to understand how the combination of DPP4 inhibition and ACE inhibition affects vasoconstriction and sympathetic activation. Understanding the hemodynamic and neurohumoral changes associated with DPP4 and ACE inhibitors has important implications for the millions of patients with T2DM who take these drugs concurrently.

ELIGIBILITY:
Inclusion Criteria:

Type 2 Diabetes Mellitus, as defined by one or more of the following,

* Hgb A1C ≥6.5%, or
* Fasting plasma glucose ≥126mg/dL, or
* Two hour plasma glucose ≥200 mg/dL following 75gr oral glucose load

For female subjects the following conditions must be met:

* Postmenopausal status for at least 1 year, or
* Status post-surgical sterilization, or
* If of childbearing potential, utilization of some form of birth control and willingness to undergo β-HCG testing prior to drug treatment and on every study day

Exclusion Criteria:

* Type 1 diabetes.
* Poorly controlled T2DM, defined as Hgb A1C>8.7%.
* Use of anti-diabetic medications other than metformin.
* Hypertension.
* Subjects who have participated in a weight-reduction program during the last 6 months and whose weight has increased or decreased more than 5 kg over the preceding 6 months.
* Pregnancy. Breast-feeding.
* Treatment with any of the following drugs: cisapride, pimozide, terfenadine, astemizol
* Clinically significant gastrointestinal impairment that could interfere with drug absorption
* Cardiovascular disease that would pose risk for the subject to participate in the study, such as: myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second- or third-degree AV block, mitral valve stenosis, or hypertrophic cardiomyopathy.
* Impaired hepatic function (aspartate amino transaminase [AST] and/or alanine amino transaminase [ALT] >2 x upper limit of normal range)
* Impaired renal function (eGFR< 60mL/min/1.73m2 as determined by the MDRD equation).
* History or presence of immunological or hematological disorders.
* History of pancreatitis or known pancreatic lesions.
* History of angioedema or cough while taking an ACE inhibitor.
* Hematocrit <35%.
* Treatment with anticoagulants.
* Growth hormone deficiency.
* Diagnosis of asthma requiring use of an inhaled β-2 agonist more than 1 time per week.
* Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
* Treatment with systemic glucocorticoids within the last 6 months.
* Treatment with lithium salts
* Ongoing tobacco use or recreational drug use.
* Treatment with any investigational drug in the 1 month preceding the study
* Mental conditions rendering the subject unable to understand the nature, scope, or possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin Then Placebo (Diabetics and Controls): Subjects in this arm will receive sitagliptin 100 mg daily. After one week of treatment, subjects will report for study day #1. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. A four week washout of medications will occur after the study day. Subjects will then receive placebo for one week followed by study day #2.
  Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Placebo Then Sitagliptin (Diabetics and Controls): Subjects in this arm will receive placebo for one week. After this, subjects will report for study day #1. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. A four week washout of medications will occur after the study day. Subjects will then receive 100 mg of sitagliptin daily for one week followed by study day #2.
  Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Sitagliptin Then Placebo: Valsartan (Controls Only): Subjects in this arm will receive sitagliptin 100 mg/d for one week as well as valsartan 160 mg/d for one week. After this subjects will report for study day #1. During the study day, subjects will be given intra-arterial neuropeptide Y. A four week washout of medication will occur after the study day. Subjects will then receive placebo/d and valsartan 160 mg/d for one week followed by study day #2.
  Sitagliptin: Subjects will receive sitagliptin 100 mg daily for 7 days prior to one of the study days.
  Placebo: Subjects will receive a placebo capsule daily for 7 days prior to one of the study days.
  Valsartan 160mg: Valsartan 160 mg/d for 7 days prior to one of the study days.
- Placebo Then Sitagliptin: Valsartan (Controls Only): Subjects in this arm will receive placebo/d for one week as well as valsartan 160 mg/d for one week. After this subjects will report for study day #1. During the study day, subjects will be given intra-arterial neuropeptide Y. A four week washout of medication will occur after the study day. Subjects will then receive sitagliptin 100mg/d and valsartan 160 mg/d for one week followed by study day #2.
  Sitagliptin: Subjects will receive sitagliptin 100 mg daily for 7 days prior to one of the study days.
  Placebo: Subjects will receive a placebo capsule daily for 7 days prior to one of the study days.
  Valsartan 160mg: Valsartan 160 mg/d for 7 days prior to one of the study days.
Period: Overall Study
Arm/Group | Sitagliptin Then Placebo (Diabetics and Controls) | Placebo Then Sitagliptin (Diabetics and Controls) | Sitagliptin Then Placebo: Valsartan (Controls Only) | Placebo Then Sitagliptin: Valsartan (Controls Only)
Started | 7 | 6 | 2 | 3
Completed | 7 | 6 | 2 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This is a crossover study with two protocols. All subjects in protocol 1 (crossover arms 1 and 2) received the same treatments, and all subjects in protocol 2 (arms 3 and 4) received the same treatments. Seven normal controls and 6 patients with diabetes completed protocol 1 (arms 1 or 2). Five normal controls completed protocol 2 (arms 3 or 4).
Groups:
- Controls Who Completed Crossover Arm 1 or 2: Healthy non-smokers Crossover arm 1 is sitagliptin then placebo Crossover arm 2 is placebo then sitagliptin
- Patients With Diabetes Who Completed Crossover Arm 1 or 2: Non-smokers with diabetes who were taking no medication or metformin only Crossover arm 1 is sitagliptin then placebo Crossover arm 2 is placebo then sitagliptin
- Controls Who Completed Crossover Arm 3 or 4: Healthy non-smokers Crossover arm 3 is sitagliptin and valsartan, then placebo and valsartan Crossover arm 4 is placebo and valsartan, then sitagliptin and valsartan
- Total: Total of all reporting groups
Arm/Group | Controls Who Completed Crossover Arm 1 or 2 | Patients With Diabetes Who Completed Crossover Arm 1 or 2 | Controls Who Completed Crossover Arm 3 or 4 | Total
Number analyzed (Participants) | 7 | 6 | 5 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (10.0) | 43.6 (6.0) | 31.4 (9.0) | 36.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 9
  Male | 3 | 3 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 6 | 4 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 6 | 5 | 18
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.9 (2.7) | 33.6 (8.7) | 25.7 (2.0) | 28.4 (6.3)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of hemoglobin] | 5.2 (0.6) | 6.6 (0.2) | 5.0 (0.2) | 5.6 (0.8)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 78.3 (12.7) | 105.7 (12.7) | 80.4 (4.4) | 88.0 (15.3)

OUTCOME MEASURES:

1. Primary Outcome: Forearm Blood Flow
Description: Forearm blood flow measured by strain gauge plethysmography in response to 1.0 nmol/min neuropeptide Y, the highest dose that all received.
Time Frame: FBF measured after 5 min of the 1 nmol/min dose of neuropeptide Y on study days 1 and 2. Study days 1 and two were separated by five weeks.
Measure: Mean (Standard Deviation); unit: mL/min/100 mL
Groups:
- Sitagliptin and Enalaprilat (Diabetics and Controls): Subjects will receive sitagliptin 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Placebo and Enalaprilat (Diabetics and Controls): Subjects will receive placebo 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Sitagliptin and Valsartan (Controls Only): Subjects in this arm will receive sitagliptin 100 mg/d for one week as well as valsartan 160 mg/d for one week. After this subjects will report for a study day. During the study day, subjects will be given intra-arterial neuropeptide Y.
- Placebo and Valsartan (Controls Only): Subjects in this arm will receive a placebo for one week as well as valsartan 160 mg/d for one week. After this subjects will report for a study day. During the study day, subjects will be given intra-arterial neuropeptide Y.
Arm/Group | Sitagliptin and Enalaprilat (Diabetics and Controls) | Placebo and Enalaprilat (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
mL/min/100 mL | 1.72 (0.93) | 2.29 (0.93) | 1.17 (0.21) | 1.63 (0.85)

2. Secondary Outcome: Arterial Norepinephrine
Description: Arterial norepinephrine concentration measured by high-performance liquid chromatography.
Time Frame: Measured at baseline (time 0) prior to the infusion of neuropeptide Y on each study day. Study days 1 and 2 were separated by five weeks.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Sitagliptin + Enalaprilat (Diabetics and Controls): Subjects will receive sitagliptin 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Placebo + Enalaprilat (Diabetics and Controls): Subjects will receive placebo 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
Arm/Group | Sitagliptin + Enalaprilat (Diabetics and Controls) | Placebo + Enalaprilat (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
pg/mL | 211.8 (81.8) | 174.7 (80.2) | 151.8 (31.3) | 125.5 (35.1)

3. Secondary Outcome: Venous Norepinephrine
Description: Venous norepinephrine concentration measured by high-performance liquid chromatography
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Sitagliptin + Enalaprilat (Diabetics and Controls) | Placebo + Enalaprilat (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
pg/mL | 250.6 (192.9) | 178.3 (85.1) | 192.6 (88.6) | 173.1 (65.5)

4. Secondary Outcome: NPY Metabolites
Description: NPY (3-36) concentration measured by micro ultra-hgih pressure liquid chromatography tandem mass spectrometry.
  NPY (3-36) is the degradation product of NPY by dipeptidyl peptidase 4. It was measured only in the diabetics studied.
Time Frame: Measured after 5 min infusion of the 1.0 nmol/min dose of neuropeptide Y on study days 1 and 2. Study days 1 and 2 were separated by five weeks.
Population: Because the purpose of measuring NPY metabolites was to assess whether sitagliptin blocks the formation of the metabolites, and because the analysis is laborious and costly, measurements were only completed in the diabetics studied.
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- Sitagliptin (Diabetics): Subjects will receive sitagliptin 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Placebo (Diabetics): Subjects will receive placebo 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
Arm/Group | Sitagliptin (Diabetics) | Placebo (Diabetics) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 6 | 6 | 0 | 0
pmol/L | 749 (562) | 1206 (1559) |  |

5. Secondary Outcome: Insulin
Description: Plasma insulin measured by radioimmunoassay.
Time Frame: Measured at baseline (time 0) of each study day prior to the infusion of neuropeptide Y. Study days 1 and 2 were separated by five weeks, a four-week washout and one-week treatment period.
Population: The comparison of sitagliptin and placebo were original to the study. Because the purpose of the sitagliptin and valsartan versus placebo and valsartan comparison was to further understand the mechanism for forearm blood flow effects it was not necessary to measure insulin in that added part of the study.
Measure: Mean (Standard Deviation); unit: microU/mL
Groups:
- Sitagliptin (Diabetics and Controls): Subjects will receive sitagliptin 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Placebo (Diabetics and Controls): Subjects will receive placebo 100 mg daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 12 | 11 | 0 | 0
microU/mL | 16.2 (10.6) | 19.6 (14.1) |  |

6. Secondary Outcome: GLP-1
Description: GLP--1 was not analyzed as subjects were studied in the fasting state.
Time Frame: Measured at baseline (time 0) of each study day prior to the infusion of neuropeptide Y. Study days were separated by five weeks, a four-week washout and one-week treatment period.
Population: GLP--1 was not analyzed as subjects were studied in the fasting state.
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Glucose
Description: Glucose was measured by the glucose oxidase method using a YSI glucose analyzer
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
mg/dL | 94.3 (16.1) | 100.3 (19.6) | 85.7 (3.4) | 88.3 (1.9)

8. Secondary Outcome: ACE Activity
Description: ACE activity was measured using a commercially available assay (Olympus AU400/AU600, Alpco Diagnotics, Salem, NH.) The lower level of detection was 15 U/L and values below the level of detection were reported at half the level of detection.
Time Frame: as for outcome 6
Population: Was not measured during the valsartan study days.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Sitagliptin + Enalaprilat (Diabetics and Controls) | Placebo + Enalaprilat (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 0 | 0
U/L | 7.5 (0) | 7.5 (0) |  |

9. Secondary Outcome: DPP4 Activity
Description: DPP4 activity was measured by detection of cleavage of a colorimetric substrate.
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: nmol/ml/min
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
nmol/ml/min | 10.97 (4.47) | 21.22 (5.36) | 17.46 (7.35) | 32.55 (5.58)

10. Secondary Outcome: Low Frequency Variability of Blood Pressure Activity
Description: Measured using the VITAL-GARD 450c monitor Ivy Biomedical Systems, Branford, CT, USA)
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm Hg2
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
mm Hg2 | 5.16 (2.54) | 5.60 (2.45) | 6.05 (4.30) | 4.27 (2.21)

11. Secondary Outcome: Arterial tPA
Description: Measured using an ELISA.
Time Frame: as for outcome 6
Population: This was measured in a few subjects. After it was determined that there was no change in net t-PA release it was not measured in the remainder.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 3 | 2 | 0 | 0
ng/mL | 0.047 (0.057) | 0.115 (0.070) |  |

12. Secondary Outcome: Venous tPA
Description: Measured using an ELISA. This was measured in a few subjects. After it was determined that there was no change in net t-PA release it was not measured in the remainder.
Time Frame: as for outcome 6
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 3 | 2 | 0 | 0
ng/mL | 0.030 (0.060) | 0.110 (0.096) |  |

13. Secondary Outcome: Mean Arterial Pressure
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
mm Hg | 79.3 (8.0) | 81.4 (6.5) | 75.4 (4.2) | 74.0 (5.7)

14. Secondary Outcome: Heart Rate
Time Frame: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
Number analyzed (Participants) | 13 | 13 | 5 | 5
beats per minute | 67.4 (11.7) | 66.0 (9.4) | 59.8 (14.3) | 60.2 (14.2)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at each study day from consent until completion of the last study day. The total duration of the study from consent to the last study day was completed ranged from six to ten weeks.
Groups:
- Placebo (Diabetics and Controls): Subjects will receive placebo daily. After one week of treatment, subjects will report for a study day. During the study day subjects will be given intra-aterial neuropeptide Y and enalaprilat. Neuropeptide Y: During the study days, neuropeptide Y will be infused through an intra-arterial line. There will be four doses of neuropeptide Y used (0.1, 0.3, 1.0, and 3.0 nmol/min) and each dose will be infused for 10 minutes.
  Enalaprilat: Ninety minutes after the last dose of neuropeptide Y, enalaprilat will be infused through the intra-arterial line at 0.33 µg/min/100mL of forearm volume. After 30 minutes, a second After 30 minutes, a second NPY at graded doses was started ten minutes after that.
- Placebo and Valsartan (Controls Only): Subjects in this arm will receive splacebo for one week as well as valsartan 160 mg/d for one week. After this subjects will report for a study day. During the study day, subjects will be given intra-arterial neuropeptide Y
Arm/Group | Sitagliptin (Diabetics and Controls) | Placebo (Diabetics and Controls) | Sitagliptin and Valsartan (Controls Only) | Placebo and Valsartan (Controls Only)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/13 | 2/13 | 0/5 | 1/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (Diabetics and Controls) (N=13) | Placebo (Diabetics and Controls) (N=13) | Sitagliptin and Valsartan (Controls Only) (N=5) | Placebo and Valsartan (Controls Only) (N=5)
Light-headedness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Includes vasovagal symptoms
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
paresthesias (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT02639637/Prot_SAP_000.pdf